CLINICAL TRIAL: NCT06140459
Title: The Evaluation of the Effectiveness of Conventional and Pulsating Toothbrushes on Oral Health of Healthy and Mentally Disabled Pediatric Patients
Brief Title: The Effectiveness of Conventional and Pulsating Toothbrushes on Mentally Disabled Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Bilim University (Other)
Responsible Party: Principal Investigator, Şafak Gür, associate professor, Antalya Bilim University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: REF: 29601
Record Dates: First submitted 2023-11-06; First posted 2023-11-20 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Periodontal Indexes
Keywords: Mentally disabled children; plaque removal; conventional toothbrush; pulsating toothbrush; plaque index

STUDY DESIGN:
Intervention Model Description: Each subject can be evaluated as its own control; the number of samples is generally less than in studies designed as comparative parallel groups. Crossover design studies ensure that each patient can use each type of toothbrush. In this study, for the results to be reliable, a crossover design was used to ensure that all participants used each brush.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Disabled children (Experimental): Special education school students
  Interventions: Device: Conventional Toothbrushes; Device: Pulsating Toothbrushes
- Healthy children (Active Comparator): Systemically healthy school children
  Interventions: Device: Conventional Toothbrushes; Device: Pulsating Toothbrushes

INTERVENTIONS:
Device: Conventional Toothbrushes — Oral-B Stages 3
Device: Pulsating Toothbrushes — Oral-B Pulsar, Colgate 360º Micro Sonic Power

SUMMARY:
Children, especially the mentally disabled, are generally incapable of obtaining an adequate oral hygiene level by manual brushing because of their lack of knowledge about oral hygiene and their limited motor skills. To handle those limited skills different designs of manual and electric toothbrushes are developed and put on the market. This study aimed to evaluate the effectiveness of pulsating toothbrushes with easy-to-use properties against conventional toothbrushes and to analyze their benefits on mentally disabled pediatric patients. 31 healthy and 31 mentally disabled children (aged between 7-12) participated in this study. The effectiveness of three different toothbrushes (Oral-B Pulsar, Colgate 360º Micro Sonic Power, Oral-B Stages 3) was investigated with a cross-over study design. DMFT, dft, modified sulcus bleeding index (MOD-SBI), approximal plaque index (API) and Green and Vermillion simplified oral hygiene index (G&V OHI-S) measurements are performed and used to evaluate the oral hygiene status.

DETAILED DESCRIPTION:
Ages between 7-12 (mean age 11.14±1.08), 31 healthy (17 girls, 14 boys) and 31 educable mentally disabled (12 girls, 19 boys) (special education school students), a total of 62 children were included in the study, following the ethics committee approval (REF: 29601).

Patient selection The children in the experimental group were educable mental disabled children (special education school students) and the control group systemically healthy children (primary school students). The children participating in the study were required not to use antibiotics, not to have received an additional plaque control application in the previous 5 months, to have at least 20 teeth in their mouths and not to receive orthodontic treatment, to have an intelligence level close to the average for disabled children, and to be capable of brushing on their own. Children in the study group were informed not to perform different oral hygiene practices such as mouthwash and dental floss during the study.

A preliminary meeting was held with the children's parents and they were informed verbally and in writing about the content of the study. For this purpose, a voluntary consent form was signed, including the content of the study, duration of participation, potential risks and problems, possible benefits for the patient, address, and telephone information of the parent and the child. One-on-one interviews were held with the children's parents, questions were asked about their general health conditions, and records were taken.

Clinical Evaluation Oral and dental examinations of children were performed with the help of a mirror and probe according to the World Health Organization criteria. If any surface of the tooth became visible in the mouth, the tooth was considered erupted. If both primary and permanent teeth were in the same tooth space at the same time, permanent teeth were included in the evaluation. DMFT values for permanent teeth and dft values for primary teeth were calculated according to the DMFT index (Decayed, Missing, and Filled Teeth Index). To determine oral hygiene, G&V Simplified Oral Hygiene Index [G&V OHI-S (Green and Vermillion Oral Hygiene Index-Simplified,1964)], Modified Sulcus Bleeding Index (MOD-SBI) and Aproximal Plaque Index (API) were used. The amount of plaque was measured by staining method from different surfaces of six teeth, two from the anterior area and four from the posterior area. At the beginning of each experimental period, children were instructed not to brush their teeth for 24 hours. Bleeding status was evaluated by applying the Modified Sulcus Bleeding Index within the clinical examination before brushing on the test day and control appointments. The plaque was stained with Mira-2-tone plaque staining solution pre and post-brushing during each examination period, and the stained plaque was shown to the child.

Each child was taught individually how to brush using the Bass Technique, first on the model and then in front of the mirror. Children were instructed to brush themselves for 2 minutes twice a day, after breakfast and in the evening before going to bed. Families were informed with written documents to follow up the brushing. To ensure the accuracy of the brushing time, 2-minute hourglasses were given to all children at the beginning of the study, and the families of disabled children were specifically warned to monitor the time. Cards prepared to mark brushings were sent to families. During the study, toothpaste was sent to the children for brushing with a single type of toothpaste (Ipana Complete 7 Care System Night-Procter & Gamble).

Three different types and brands of commercially available toothbrushes (two with pulsating features and one conventional) were used in the study. The three toothbrushes were Oral-B Pulsar (Procter&Gamble) (No:35), Colgate 360º Micro Sonic Power (Colgate-Palmolive), and Oral-B Stages 3 (Procter&Gamble).

Application Procedure Parents ensured that the children did not brush their teeth 24 hours before starting the study. The children included in the study were examined at their schools. Decayed, filled, missing, and existing teeth were detected and recorded in the oral follow-up form. Each child was taught individually how to brush using the Bass Technique, first on the model and then in front of the mirror. On the first day of the test period, Modified Sulcus Bleeding Index (MOD-SBI), approximal plaque index (API), and Green and Vermillion oral hygiene index (G&V OHI-S) were measured. For Green and Vermilion oral hygiene measurement, 2 drops of Mira-2-Ton plaque staining solution were used, and with the help of a brush it was applied to the teeth. The children rinsed their mouths with water for 30 seconds and the stained surface areas were evaluated after one minute. The results were recorded in the charts on the oral follow-up form. Then, group 1 toothbrush (Oral-B Pulsar) and toothpaste were given and the child was allowed to brush on his/her own for 2 minutes. 1 minute after brushing, the teeth determined in Green and Vermillion oral hygiene index (G&V OHI-S) were repainted with Mira-2-Ton plaque staining solution. The child was asked to rinse his/her mouth with water for 30 seconds. The stained surfaces were examined and plaque levels were recorded on the forms. The first group of toothbrushes, one toothpaste, a brushing tracking card, an hourglass, and a parent information letter were sent to the children's homes. For a month, the children used the toothpaste sent with the 1st group toothbrush, twice a day (after breakfast in the morning, before going to bed in the evening) at home, on their own, under their parents' control that they were brushing and marking it on the cards. At the end of one month, the children were asked to bring their toothbrushes and follow-up cards to school with them and not to brush for 24 hours before. Intraoral examinations of the children (soft and hard tissues, lips, tongue, sublingual area, inner parts of the cheeks, hard and soft palate, and buccal mucosa folds were evaluated), and caries were detected and marked on the oral follow-up form), Modified Sulcus Bleeding Index (MOD-SBI), approximal plaque index (API), and Green and Vermillion oral hygiene index (G&V OHI-S) were measured. Measurements were recorded on charts. Then, brushing was done and Green and Vermillion oral hygiene index (G&V OHI-S) was repeated post-brushing. The children's toothbrushes were taken back, a break was given for a month, and they were asked to brush with a small-headed, simple-designed manual toothbrush that was not included in the study, in order for the children to return to their old brushing habits. After a one-month break, the applications were continued with the 2nd (Colgate 360º Micro Sonic Battery-Powered Toothbrush) and 3rd (Oral-B Stages) toothbrushes, respectively, following the same procedures. The study ended in a total of five months, with an experimental period in which each participant used all three brushes for one month and a one-month interim period between each brush for the children to return to their old habits.

ELIGIBILITY:
Inclusion Criteria:

* not use antibiotics
* not to have received an additional plaque control application in the previous 5 months
* have at least 20 teeth in their mouths
* not to receive orthodontic treatment
* For Group 1 to have an intelligence level close to the average for disabled children
* For Group 2 systemically healthy
* to be capable of brushing on their own

Exclusion Criteria:

* non-cooperative

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2008-10-01 (Actual); Primary Completion 2009-03-31 (Actual); Study Completion 2009-03-31 (Actual)

PRIMARY OUTCOMES:
Modified Sulcus Bleeding Index (MOD-SBI) | First visit, first month, third month, fifth month
  In control with a periodontal probe; It was determined whether there was bleeding in the oral gums of the 1st and 3rd half jaws and in the facial side gums of the 2nd and 4th half jaws. The status was charted as Yes (+) in the presence of bleeding and No (-) in the absence of bleeding. The result was calculated as a percentage.
Approximal plaque index (API) | First visit, first month, third month, fifth month
  Half jaws numbered 1 and 3 were evaluated from their oral surfaces, and semi jaws numbered 2 and 4 were evaluated from their facial surfaces. Whether there is only plaque or not is marked on the diagram as Yes (+), No (-). The plaque index value was calculated as a percentage (%).
Green and Vermillion oral hygiene index (G&V OHI-S) | first visit pre-brushing, first visit post-brushing, first month pre-brushing, first month post-brushing, , third month pre-brushing, third month post-brushing, fifth month pre-brushing, fifth month post-brushing
  For Green and Vermilion oral hygiene measurement, 2 drops of Mira-2-Ton plaque staining solution are dropped into plastic disposable cups and with the help of a brush, it was applied to the teeth. The child's mouth was rinsed with water for 30 seconds and the stained surface areas were evaluated after one minute. Measurements were made from the buccal surfaces of teeth 16 and 26, the lingual surfaces of teeth 36 and 46, and the labial surfaces of teeth 11 and 31. The amount of plaque was graded with 4 separate scores from 0 to 3, depending on the size of the surface area stained with the staining solution. The index was calculated by dividing the total values by the number of surfaces.

CONTACTS AND LOCATIONS:
Overall Officials: Işın Ulukapı, Prof., Study Director — Okan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou N, Wong HM, McGrath C. Oral health and associated factors among preschool children with special healthcare needs. Oral Dis. 2019 May;25(4):1221-1228. doi: 10.1111/odi.13057. Epub 2019 Feb 21. PMID 30725497
- [Background] Petrukhina NB, Boriskina OA, Shevlyakov DI. [Clinical analysis of the cleaning effectiveness of toothbrushes of various types in children aged 6-15 years after a single brushing]. Stomatologiia (Mosk). 2021;100(6):76-81. doi: 10.17116/stomat202110006176. Russian. PMID 34953193
- [Background] Zhou N, Wong HM, McGrath C. The Impact of Adaptive Functioning and Oral Hygiene Practices on Observed Tooth-Brushing Performance Among Preschool Children with Special Health Care Needs. Matern Child Health J. 2019 Dec;23(12):1587-1594. doi: 10.1007/s10995-019-02813-5. PMID 31552578
- [Background] Dogan MC, Alacam A, Asici N, Odabas M, Seydaoglu G. Clinical evaluation of the plaque-removing ability of three different toothbrushes in a mentally disabled group. Acta Odontol Scand. 2004 Dec;62(6):350-4. doi: 10.1080/00016350410010054. PMID 15848980
- [Background] Escribano Hernandez A, Hernandez Corral T, Ruiz-Martin E, Porteros Sanchez JA. Results of a dental care protocol for mentally handicapped patients set in a primary health care area in Spain. Med Oral Patol Oral Cir Bucal. 2007 Nov 1;12(7):E492-5. PMID 17978772
- [Background] Biesbrock AR, Bartizek RD, Walters PA. Improved plaque removal efficacy with a new manual toothbrush. J Contemp Dent Pract. 2008 May 1;9(4):1-8. PMID 18473021